CLINICAL TRIAL: NCT07175779
Title: Effect of Teleconsultation Compared to Face-to-Face Evaluation on Perioperative Respiratory Events in Pediatric Adenotonsillectomy: A Randomized Non Inferiority Trial
Brief Title: Teleconsultation vs Face-to-Face Evaluation for Perioperative Respiratory Events in Pediatric Adenotonsillectomy
Acronym: Teleped
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Saporito (Other)
Responsible Party: Sponsor-Investigator, Andrea Saporito, Prof. Dr. med., Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TELEPED-2025
Record Dates: First submitted 2025-08-04; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Adenotonsillar Hypertrophy
Keywords: Anesthesia Consultation; Face-to-Face Visit; Remote consultation; Patient anxiety; Patient Satisfaction; Lost Work Time; Distance Traveled; Virtual Care; Digital Health; Telemedicine; Perioperative Care; Perioperative respiratory adverse events (PRAE); Adenotonsillectomy; Tonsillectomy
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-Face Preanesthesia Consultation (Active Comparator): In-person preoperative anesthesia consultation
  Interventions: Other: Face-to-Face Preanesthesia Consultation
- Telemedicine Preanesthesia Consultation (Active Comparator): Preoperative anesthesia teleconsultation via secure video platform
  Interventions: Other: Telemedicine Preanestehsia Consultation

INTERVENTIONS:
Other: Face-to-Face Preanesthesia Consultation — Participants receive a standard preoperative anesthesia consultation in person at the hospital
  Arms: Face-to-Face Preanesthesia Consultation
Other: Telemedicine Preanestehsia Consultation — Participants receive a preoperative anesthesia consultation remotely via video conferencing using a secure telemedicine platform.
  Arms: Telemedicine Preanesthesia Consultation

SUMMARY:
The goal of this clinical trial is to assess whether preoperative anesthesia teleconsultation is at least equivalent to in-person consultation in preventing perioperative respiratory adverse events (such temporary reduction in oxygen levels in the blood) in the operating room and in the first 24 hours after the surgery in pediatric adenotonsillectomy.

Researchers will compare the teleconsultation to in-person consultation to see if there is a difference in the frequency of respiratory adverse events in the operating room and during the first 24 hours after adenotonsillectomy.

Participants will:

- undergo a traditional in-person anesthesiology consultation scheduled at the hospital or a online preoperative anesthesiology teleconsultation.

DETAILED DESCRIPTION:
Adenotonsillectomy is one of the most common surgical procedures in children, and perioperative respiratory adverse events (PRAEs) such as desaturation, laryngospasm, or bronchospasm represent a frequent source of morbidity. Careful preoperative anesthesiology evaluation is crucial to identify risk factors and to implement preventive strategies. Traditionally, this assessment is performed during an in-person consultation at the hospital. However, telemedicine has recently emerged as a potential alternative, offering advantages in terms of accessibility, cost-effectiveness, and reduced burden on families, especially when hospital access is challenging.

The primary aim of this randomized non-inferiority clinical trial is to determine whether a preoperative anesthesia teleconsultation is at least equivalent to a face-to-face consultation in preventing perioperative respiratory adverse events in pediatric patients undergoing adenotonsillectomy.

This trial will provide high-quality evidence regarding the safety and effectiveness of teleconsultation as a preoperative assessment strategy in pediatric surgery. If non-inferiority is demonstrated, the study could support the broader implementation of telemedicine in perioperative care pathways, potentially improving accessibility and reducing healthcare costs without compromising patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (up to 16 years of age) undergoing elective tonsillectomy or adenotonsillectomy
* ASA (American Society of Anesthesiologists) physical status I to III,
* Patients who have a parent or legal guardian able and willing to provide informed consent.

Exclusion Criteria:

* Parent or guardian unable or unwilling to provide informed consent,
* Refusal to participate by parent/guardian,
* Patients with contraindications to general anesthesia,
* Known allergy to any drugs used in the anesthetic protocol.
* Potential difficult airway,
* Poorly controlled chronic illness (e.g. asthma),
* Cardiac disease ,
* Genetic disorder,
* Haemoglobinopathy, anemia or clotting problem,
* Complex physical disability,
* Request from the patient or carer

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of perioperative respiratory adverse events (PRAE) | Intraoperatively
  including desaturation, airway obstruction, laryngospasm, bronchospasm, and wheezing, recorded intraoperatively and up to 24 hours postoperatively.
Incidence of PRAE (perioperative respiratory adverse events) | up to 24 hours postoperatively
  including desaturation, airway obstruction, laryngospasm, bronchospasm, and wheezing

SECONDARY OUTCOMES:
Consultation duration | Day of consultation
  Time in minutes from the start to the end of the preoperative anesthesia consultation (either in-person or via telemedicine). The duration will be recorded by the anesthesiologist at the end of each consultation
preoperative assessment adequacy | Day of surgery
  Day-of-surgery cancellation rate
Preoperative anxiety in parents | Day of surgery
  Parental anxiety will be assessed using the Amsterdam Preoperative Anxiety and Information Scale (APAIS), a validated questionnaire with six self-reported items rated on a 5-point Likert scale (1 = not at all to 5 = extremely). Higher scores indicate greater anxiety and information need.
Preoperative anxiety in paediatric patients aged 8 years and older | Day of surgery
  For children aged 8 years and older, the Visual Analogue Scale for Anxiety (VAS-A) will be used, a self-reported 10-cm visual analogue with facial expressions ranging from "very distressed" to "very happy." Scores are recorded from 0 to 10, with higher scores indicating greater anxiety
Preoperative anxiety in paediatric patients younger than 8 years | Day of surgery
  For children younger than 8 years, the modified Yale Preoperative Anxiety Scale - Short Form (mYPAS-SF) will be used, which evaluates five behavioral domains (activity, vocalization, emotional expressivity, state of arousal, and interaction with parents) on a 1-5 scale. Higher scores indicate greater observable anxiety
Environmental impact | Day of consultation (up to 24 hours post-consultation)
  estimated in terms of CO₂ emissions potentially avoided based on the number of kilometers not traveled by car
Parental satisfaction | Day of consultation (up to 24 hours post-consultation)
  assessed using a Numeric Rating Scale (NRS) ranging from 1 (not satisfied at all) to 10 (extremely satisfied)
travel costs | Day of consultation (up to 24 hours post-consultation)
  Direct travel-related expenses (e.g., fuel, public transport, parking) incurred by the family to attend the preoperative anesthesia consultation. Costs will be self-reported by parents using a structured questionnaire, expressed in local currency
Time off work for parents | Day of consultation (up to 24 hours post-consultation)
  Number of working hours lost by parents or guardians in order to attend the preoperative anesthesia consultation. Data will be self-reported in a post-consultation questionnaire, expressed in hours

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Saporito, MD, Prof., Study Director — Ente Ospedaliero Cantonale, Servizio di Anestesiologia
Locations (1):
- Ospedale Regionale Bellinzona e Valli, Bellinzona, Canton Ticino, Switzerland